CLINICAL TRIAL: NCT07167472
Title: Investigation of the Effects of Shoe Heel Heights on Gait Parameters in Healthy Individuals
Brief Title: Effects of Heel Height on Gait Parameters
Status: Recruiting | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, Principal Investigator, Hacettepe University
Other Study IDs: Heel Height
Record Dates: First submitted 2025-08-26; First posted 2025-09-11 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Gait; Locomotion

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults with Normal BMI: Healthy volunteers aged 18-35 years with normal BMI, assessed under three walking conditions (barefoot, 2 cm heel, 6 cm heel).

SUMMARY:
This observational study aims to investigate the effects of different shoe heel heights on gait parameters and pelvic kinematics in healthy adults aged 18-35 years. Each participant will be assessed under three conditions: barefoot, wearing shoes with 2 cm heels, and wearing shoes with 6 cm heels. Spatiotemporal gait parameters (gait speed, cadence, step length, stance and swing phase percentages, gait cycle duration) and pelvic kinematics (tilt, obliquity, rotation symmetry) will be measured using the BTS-G wireless sensor system. The study seeks to identify biomechanical differences associated with heel height and to provide data that may contribute to shoe design and individualized rehabilitation strategies.

DETAILED DESCRIPTION:
This prospective observational crossover study will be conducted at Yuksek Ihtisas University. Healthy volunteers aged 18-35 years with normal body mass index and no musculoskeletal or neurological conditions affecting gait will be recruited. Participants will be excluded if they use orthotics, have had lower extremity injuries or surgery in the past 6 months, or have chronic ankle instability.

Each participant will undergo gait assessments under three randomized shoe conditions: barefoot, wearing shoes with 2 cm heels, and wearing shoes with 6 cm heels. A BTS-G (BTS Bioengineering, Italy) wireless inertial sensor will be placed at the L4-L5 level to record spatiotemporal gait parameters and pelvic kinematics in the anteroposterior, mediolateral, and vertical axes during a 10-meter walk at a self-selected speed. The primary variables will include gait speed, cadence, stride length, stance and swing phase percentages, and gait cycle duration. Pelvic tilt, obliquity, and rotation symmetry indices will also be evaluated

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, aged 18-35 years
* Body Mass Index (BMI) within normal range (18.5-24.9 kg/m²)
* Foot structure compatible with shoe size
* Voluntarily agrees to participate and provide informed consent.

Exclusion Criteria:

* Use of orthotics or insoles
* History of musculoskeletal conditions affecting gait
* Lower extremity injury or surgery within the past 6 months
* Chronic ankle instability
* Receiving treatment related to the lower extremities within the past 6 months

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adult volunteers aged 18-35 years with normal BMI (18.5-24.9 kg/m²) and no musculoskeletal or neurological conditions affecting gait. Participants will be assessed under three heel height conditions (barefoot, 2 cm heel, 6 cm heel) to examine the impact on gait spatiotemporal parameters and pelvic kinematics.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Speed Across Heel Height Conditions | At baseline session (single day, immediate assessment across three shoe conditions)
  Self-selected walking speed (meters/second (m/s)) measured with BTS-G wireless sensor during a 10-meter walk under three conditions: barefoot, 2 cm heel, and 6 cm heel.
Change in Cadence Across Heel Height Conditions | At baseline session (single day, immediate assessment across three shoe conditions)
  Step cadence (steps/min) assessed with BTS-G sensor under barefoot, 2 cm heel, and 6 cm heel conditions.
Change in Stride Length Across Heel Height Conditions | At baseline session (single day, immediate assessment across three shoe conditions)
  Stride length (cm) obtained using BTS-G sensor during walking trials under barefoot, 2 cm heel, and 6 cm heel conditions.
Change in Stance and Swing Phase Percentages | At baseline session (single day, immediate assessment across three shoe conditions)
  Percentage of stance (%) and swing phases (%) of the gait cycle calculated by BTS-G sensor under barefoot, 2 cm heel, and 6 cm heel conditions.
Change in Pelvic Kinematics-pelvic tilt | At baseline session (single day, immediate assessment across three shoe conditions)
  Pelvic tilt recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.
Change in Pelvic Kinematics-pelvic obliquity | At baseline session (single day, immediate assessment across three shoe conditions)
  Pelvic obliquity recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.
Change in Pelvic Kinematics- pelvic rotation | At baseline session (single day, immediate assessment across three shoe conditions)
  Pelvic rotation recorded with BTS-G sensor across barefoot, 2 cm heel, and 6 cm heel conditions. It will be recorded as a degree.
Body Mass Index (BMI) | Baseline (single assessment before gait analysis).
  ody weight and height will be measured, and BMI will be calculated as weight (kg) divided by height squared (m²). Recorded at baseline for all participants. Its unit is kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Mıyaser Medıne Gok, Principal Investigator — Yuksek Ihtisas University; Busra Kalkan Balak, Study Director — Yuksek Ihtisas University; Gungor Beyza Ozvar Senoz, Principal Investigator — Yuksek Ihtisas University; Sevılay Seda Bas, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No